CLINICAL TRIAL: NCT02306512
Title: Mohs Micrographic Surgery for Primary Cutaneous Malignant Melanoma In Situ Using Immunofluorescence
Brief Title: Mohs and Immunofluorescence for Malignant Melanoma In Situ
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the University of Miami
Sponsor: University of Miami (Other)
Collaborators: University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, Vice Chairman Department of Dermatology & Cutaneous Surgery, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140210; 0000000 (Other Grant/Funding Number: Sylvester Cancer Comprenhensive Center)
Record Dates: First submitted 2014-08-27; First posted 2014-12-03 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Lentigo Maligna; Melanoma In Situ
Keywords: Melanoma In Situ; Lentigo Maligna; Confocal Microscopy; Direct Immunofluorescence
MeSH Terms: conditions — Hutchinson's Melanotic Freckle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard vs. IF MART-1 (Active Comparator): Samples removed with MMS within the first 3 mm margin from the tumor will be the first section. They will be processed as a conventional H&E frozen section and section stained with IHC MART-1. Samples removed with MMS within 3-6 mm from tumor margin will be the second section. They will be processed with fluorescent MART-1 antibodies. Based on the pre-defined characteristics MMS surgeon will evaluate each MART-1 immunofluorescent section as "no evident melanoma" or "possible melanoma" or "present melanoma". Dermatopathologist will secondarily review each section scoring them in the same manner. If standard H&E, IHC, or immunofluorescence is recorded as "present melanoma" or "possible melanoma" a third section from 6-9mm will have the same procedure described before.
  Interventions: Procedure: H&E; Procedure: IHC MART-1; Procedure: IF MART-1
- IF MART-1 versus IF cocktail (Active Comparator): In the second arm of the study, assuming that immunofluorescence with MART-1 proves to be superior or at least equivocal to regular MART-1 IHC, the same method will be applied, but the control sections will be stained with fluorescent MART-1 antibodies and compared to a section stained with a cocktail of fluorescent melanocytic antibodies.
  Interventions: Procedure: IF MART-1; Procedure: IF cocktail

INTERVENTIONS:
Procedure: H&E — Sample will be stained with H&E according to standard procedures
  Arms: Standard vs. IF MART-1
Procedure: IHC MART-1 — Samples will be stained with immunohistochemistry antibody: MART-1 according to standard procedures.
  Arms: Standard vs. IF MART-1
Procedure: IF MART-1 — Samples will be stained with immunofluorescence antibody: MART-1 according to standard procedures.
Procedure: IF cocktail — The fluorescent primary antibodies may include HMB-45, SOX10, Ki-67 and MART-1. However other markers will be considered to make the most visually remarkable cocktail; these may include S-100, MiTF, lamin and nestin. Primary antibodies will be tagged with secondary antibodies labeled with fluorescent signals. A fluorescent organelle stain and/or 4',6-diamidine-2-phenylindol (DAPI) may also be used to enhance cellular architecture.
  Arms: IF MART-1 versus IF cocktail

SUMMARY:
The purpose of this study is to determine if immunofluorescence (IF) can effectively identify features of malignant melanoma in situ, on sun-damaged skin, in the setting of Mohs Micrographic Surgery.

DETAILED DESCRIPTION:
The aim of this study is to

1. Determine the feasibility of using melanocytic markers such as Melanoma antigen recognized by T cells 1 (MART-1) with fluorescence to clear surgical margins when compared to conventional MART-1 immunohistochemistry (IHC) in the setting of MMS for LM (lentigo maligna type melanoma in situ).
2. Compare the use of a cocktail of immunofluorescent markers such as, but not limited to, Sex-determining Region Y (SRY)-box 10 (SOX10), human melanoma black 45 (HMB-45), and Kiel-67 (Ki-67) to sections only stained with fluorescent MART-1 alone.
3. Explore the value of using other combinations of immunofluorescent markers such as S-100 with Microphthalmia-associated transcription factor (MiTF), Nestin with Ki-67, and HMB-45 with Lamin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race and at least 18 years of age
2. Patient with biopsied proven Lentigo maligna (LM) in situ
3. Patient meets criteria for Mohs Micrographic Surgery (MMS)

   1. The cancer is large
   2. The edges of the cancer (clinical margins) cannot be clearly defined
   3. Prior treatment has failed, i.e. recurrent tumor
   4. The cancer is located in a cosmetically sensitive or functionally critical area of the body (such as eyelids, nose, ears, lips, fingers, toes, and genitals)
   5. The histologic pattern of the cancer is aggressive
   6. The patient is immunosuppressed
4. Patient with biopsied proven LM in situ located on an anatomic areas appropriate for MMS:

   1. Area H: ''Mask areas'' of face (central face, eyelids [including inner/outer canthi], eyebrows, nose, lips [cutaneous/mucosal/vermillion], chin, ear and periauricular skin/sulci, temple), genitalia (including perineal and perianal), hands, feet, nail units, ankles, and nipples/areola.
   2. Area M: Cheeks, forehead, scalp, neck, jawline, pretibial surface.
   3. Area L: Trunk and extremities (excluding pretibial surface, hands, feet, nail units, and ankles).
5. Patient able to tolerate surgery
6. Patient is able to comply with appointments including follow-up appointments
7. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients under the age of 18
2. Patient does not meet criteria for MMS or has LM located in areas that are not accessible with MMS
3. Patient with previously diagnosed invasive LM
4. Patients unable to comply with follow-up
5. Adults unable to consent
6. Pregnant women
7. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
IF MART-1 versus Standard H&E and IHC MART-1 | End of Mohs Surgery, approximately up to 24 hours
  Comparison of the number of high power fields containing melanoma in situ with IF Mart-1 vs. standard H&E and IHC Mart-1 when evaluating margins during MMS

SECONDARY OUTCOMES:
IF cocktail vs IF MART-1 alone | End of Mohs Surgery, approximately up to 24 hours
  Comparison of the number of high-power fields containing melanoma in situ with IF cocktail vs. IF Mart-1 alone when evaluating margins during MMS

CONTACTS AND LOCATIONS:
Overall Officials: James Grichnik, MD, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Sylvester Comprenhensive Cancer Center, Miami, Florida
  - University of Miami Hospital dermatology clinics, Miami, Florida